CLINICAL TRIAL: NCT02134509
Title: Smartphone Application for Smoking Cessation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yale University (Other)
Collaborators: American Heart Association (Other); National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 1301011337; 2K12DA000167-26 (NIH)
Record Dates: First submitted 2014-05-07; First posted 2014-05-09 (Estimated); Last update posted 2020-04-16 (Actual); Status verified 2020-01

CONDITIONS: Smoking
Keywords: Cigarette smoking
MeSH Terms: conditions — Smoking; Cigarette Smoking

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Experimental App (Experimental): This is a 3-week smartphone-based training program that trains behavioral strategies for smoking cessation by helping smokers self-monitor their smoking habits, recognize when and how often they smoke, identify triggers for smoking, and learn methods to become more mindful of triggers, to quit smoking with a target quit date of 3 weeks.
  Interventions: Behavioral: Experimental App
- Active comparator app (Active Comparator): This is a 3-week smartphone application for smoking cessation in which smokers self-monitor their smoking habits, mood, and experience, to quit smoking with a target quit date of 3 weeks.
  Interventions: Behavioral: Active Comparator App

INTERVENTIONS:
Behavioral: Experimental App — It is comprised of twenty-two modules of 10-15 minutes each, designed to teach behavioral strategies for smoking cessation using psychoeducation-based audio and videos, animations to reinforce key concepts, and in vivo exercises. In addition, 5 bonus modules become available upon completion of earlier modules; these may be accessed for additional practices to bolster other modules
  Arms: Experimental App
Behavioral: Active Comparator App — It is comprised of 6 prompts per day asking individuals about their experience, behavior, and smoking habits, for 22-days.
  Arms: Active comparator app

SUMMARY:
The purpose of this study is to test the effectiveness of a smartphone application for smoking cessation in smokers ages 18 to 65 years.

DETAILED DESCRIPTION:
In this randomized control trial, subjects will be randomly assigned to receive one of two treatments: (1) a standard smartphone application to support smokers working to become quit-free, or (2) the tested intervention, an app that trains behavioral strategies for smoking cessation. The primary endpoint of interest will be 1-week point prevalence abstinence at end of treatment, and at 3 and 6 months follow-up for individuals.

ELIGIBILITY:
Inclusion Criteria:

* Smoke 5+ cigarettes/day
* < 3 months abstinence in the past year
* Have a smartphone
* Score greater than or equal to 8 of 10 on the Contemplation Ladder (Biener & Abrams, 1991)

Exclusion Criteria:

* None

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 511 (Actual)
Dates: Start 2014-10; Primary Completion 2016-03 (Actual); Study Completion 2016-06 (Actual)

PRIMARY OUTCOMES:
Point prevalence abstinence at 6 months | 6 months after beginning treatment
  Subjects will be assessed for smoking abstinence at a 6-month follow-up.

SECONDARY OUTCOMES:
Point prevalence abstinence at 3 months | 3 months after beginning treatment
  Subjects will be assessed for smoking abstinence at a 3-month follow-up.

CONTACTS AND LOCATIONS:
Overall Officials: Kathleen A Garrison, PhD, Principal Investigator — Yale University
Locations (1):
- Yale University School of Medicine, New Haven, Connecticut, United States

REFERENCES:
- [Derived] Jackson S, Brown J, Norris E, Livingstone-Banks J, Hayes E, Lindson N. Mindfulness for smoking cessation. Cochrane Database Syst Rev. 2022 Apr 14;4(4):CD013696. doi: 10.1002/14651858.CD013696.pub2. PMID 35420700
- [Derived] Sala M, Roos CR, Brewer JA, Garrison KA. Awareness, affect, and craving during smoking cessation: An experience sampling study. Health Psychol. 2021 Sep;40(9):578-586. doi: 10.1037/hea0001105. Epub 2021 Sep 27. PMID 34570534
- [Derived] Garrison KA, Pal P, O'Malley SS, Pittman BP, Gueorguieva R, Rojiani R, Scheinost D, Dallery J, Brewer JA. Craving to Quit: A Randomized Controlled Trial of Smartphone App-Based Mindfulness Training for Smoking Cessation. Nicotine Tob Res. 2020 Mar 16;22(3):324-331. doi: 10.1093/ntr/nty126. PMID 29917096
- [Derived] Garrison KA, Pal P, Rojiani R, Dallery J, O'Malley SS, Brewer JA. A randomized controlled trial of smartphone-based mindfulness training for smoking cessation: a study protocol. BMC Psychiatry. 2015 Apr 14;15:83. doi: 10.1186/s12888-015-0468-z. PMID 25884648